CLINICAL TRIAL: NCT06649864
Title: A Phase I Study of Autologous Adipose-derived Mesenchymal Stromal Cells in Preventing Biliary Complications After Living Donor Liver Transplant
Brief Title: Adipose-Derived Mesenchymal Stem Cell for Preventing Biliary Complications
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Julie K. Heimbach, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-001649
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Liver Transplant; Complications; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liver Transplant (Experimental): Subjects with liver disease with planned living donor liver transplantation
  Interventions: Drug: Autologous adipose derived mesenchymal stromal cells (AMSC)

INTERVENTIONS:
Drug: Autologous adipose derived mesenchymal stromal cells (AMSC) — Adipose derived autologous mesenchymal stromal cells; [~500,000 cells/cm2] will be applied once to the biliary anastomosis using approximately 3-5 million cells in 5ml Lactated Ringer solution.

SUMMARY:
The purpose of this study is to assess the safety of autologous Adipose-Derived Mesenchymal Stem Cell for use in End-Stage Liver Disease patients undergoing the creation of a duct-to-duct anastomosis during Living Donor Liver Transplantation.

ELIGIBILITY:
Inclusion Criteria

* Listed for liver transplantation
* Non-pediatric patients with a planned LDLT
* Ability to communicate with investigative staff
* Competence to give written informed consent
* Ability to comply with the entire study procedure
* All sexes and genders will be eligible for the study

Exclusion Criteria

* Planned deceased donor liver transplantation
* Uncontrolled / unresolved local or systemic infection
* Body mass index > 40
* Planned pancreaticoduodenectomy or sleeve gastrectomy
* Anticipation of 3 biliary anastomoses (we will include those anticipated to have 1 or 2 biliary anastomoses as detailed below)
* Pregnancy or breastfeeding
* Non-liver cancers (we will include certain patients with primary liver cancer as detailed below)
* Treatment with any investigational drug / device within 60 days prior to study entry
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of AMSCs
* Patients who are employees or relatives of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Side effects | 24 months
  Number of subjects to experience systemic symptoms, irritation, inflammation, infections or biliary obstructions

SECONDARY OUTCOMES:
Biliary complications | 24 months
  Number of subjects to develop biliary complications of strictures or leaks

CONTACTS AND LOCATIONS:
Overall Officials: Julie Heimbach, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No